CLINICAL TRIAL: NCT03829618
Title: Lidocaine Administration During Flexible Bronchoscopy and Endobronchial Ultrasound
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: COVID lack of cases/recruitment
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Jennifer Toth, Professor of Medicine and Surgery, Director of Interventional Pulmonology, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00009727
Record Dates: First submitted 2019-01-24; First posted 2019-02-04 (Actual); Results first posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-09

CONDITIONS: Bronchiectasis Adult; Mediastinal Lymphadenopathy; Pneumonia; Chest--Diseases; Infiltrates; Bronchopulmonary Disease; Cancer, Lung
MeSH Terms: conditions — Pneumonia; Lung Neoplasms | interventions — Lidocaine; Nebulizers and Vaporizers

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Topical Lidocaine (Active Comparator): 16 ml of 1% lidocaine sprayed in 4 ml aliquots to vocal cords, midtrachea, left main stem bronchus and right main stem bronchus.
  Interventions: Drug: Topical lidocaine
- Nebuliser Solution (Active Comparator): 2% lidocaine dosed at 2mg/kg with max dose of 160mg nebulized via jet nebulizer in operating room over ten minutes.
  Interventions: Drug: Nebuliser solution
- Nebuliser Suspension (Active Comparator): 2% lidocaine dosed at 2mg/kg with max dose of 160mg nebulized via vibrating mesh nebulizer in operating room over ten minutes.
  Interventions: Drug: Nebuliser Suspension

INTERVENTIONS:
Drug: Topical lidocaine — 1% lidocaine topically applied in 4 mL aliquots
  Other Names: Topical
  Arms: Topical Lidocaine
Drug: Nebuliser solution — 2% lidocaine dose at 2 mg/kg (max 160 mg) applied via jet nebulizer
  Other Names: Nebulizer
  Arms: Nebuliser Solution
Drug: Nebuliser Suspension — 2% lidocaine dosed at 2 mg/kg (max 160 mg) applied via vibrating mesh nebulizer
  Other Names: Atomizer
  Arms: Nebuliser Suspension

SUMMARY:
The purpose of this study is to assess if there is decrease in cough during flexible bronchoscopy and endobronchial ultrasound when different modes of lidocaine administration are used. The modes of administration being evaluated are topical, nebulized and atomized.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mediastinal and/or hilar lymphadenopathy requiring endobronchial ultrasound evaluation and transbronchial needle aspiration.
* Diagnosis of pulmonary disease requiring flexible bronchoscopy
* Greater than 18 years of age.

Exclusion Criteria:

* Any intervention beyond flexible bronchoscopy and endobronchial ultrasound
* Inability to tolerate bronchoscopy.
* Patients that receive paralytics.
* Patients with neuromuscular diseases.
* Inability to consent for procedures.
* Allergies to lidocaine or any other drugs used in protocol.
* Existing renal insufficiency or liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Toth, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Penn State Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Madan K, Biswal SK, Mittal S, Hadda V, Mohan A, Khilnani GC, Pandey RM, Guleria R. 1% Versus 2% Lignocaine for Airway Anesthesia in Flexible Bronchoscopy Without Lignocaine Nebulization (LIFE): A Randomized Controlled Trial. J Bronchology Interv Pulmonol. 2018 Apr;25(2):103-110. doi: 10.1097/LBR.0000000000000458. PMID 29346249
- [Background] Stolz D, Chhajed PN, Leuppi J, Pflimlin E, Tamm M. Nebulized lidocaine for flexible bronchoscopy: a randomized, double-blind, placebo-controlled trial. Chest. 2005 Sep;128(3):1756-60. doi: 10.1378/chest.128.3.1756. PMID 16162784
- [Background] Wahidi MM, Jain P, Jantz M, Lee P, Mackensen GB, Barbour SY, Lamb C, Silvestri GA. American College of Chest Physicians consensus statement on the use of topical anesthesia, analgesia, and sedation during flexible bronchoscopy in adult patients. Chest. 2011 Nov;140(5):1342-1350. doi: 10.1378/chest.10-3361. PMID 22045879
- [Background] Dreher M, Cornelissen CG, Reddemann MA, Muller A, Hubel C, Muller T. Nebulized versus Standard Local Application of Lidocaine during Flexible Bronchoscopy: A Randomized Controlled Trial. Respiration. 2016;92(4):266-273. doi: 10.1159/000449135. Epub 2016 Sep 10. PMID 27614989
- [Result] Amini S, Peiman S, Khatuni M, Ghalamkari M, Rahimi B. The Effect of Dextromethorphan Premedication on Cough and Patient Tolerance During Flexible Bronchoscopy: A Randomized, Double-blind, Placebo-controlled Trial. J Bronchology Interv Pulmonol. 2017 Oct;24(4):263-267. doi: 10.1097/LBR.0000000000000385. PMID 28891835

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants will be Identified from pool of patients who will already be undergoing with planned flexible bronchoscopy and/or endobronchial ultrasound by an interventional pulmonologist in the operating room setting. They will be identified by review of the operating room schedule and through the interventional pulmonology clinic.
Groups:
- Atomizer Solution: 2% lidocaine dosed at 2mg/kg with max dose of 160mg nebulized via vibrating mesh nebulizer in operating room over ten minutes.
  Nebuliser Suspension: 2% lidocaine dosed at 2 mg/kg (max 160 mg) applied via vibrating mesh nebulizer
Period: Overall Study
Arm/Group | Topical Lidocaine | Nebuliser Solution | Atomizer Solution
Started | 15 | 7 | 7
Completed | 15 | 7 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Topical Lidocaine | Nebuliser Solution | Atomizer Solution | Total
Number analyzed (Participants) | 15 | 7 | 7 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.80 (12.81) | 55.57 (16.83) | 57.43 (14.77) | 61.83 (14.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 4 | 14
  Male | 8 | 4 | 3 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 15 | 6 | 6 | 27
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 15 | 7 | 7 | 29
BMI [Mean (Standard Deviation); unit: kg/m^2] | 30.19 (6.93) | 29.39 (4.84) | 28.53 (8.23) | 29.59 (6.63)
Smoking History [Count of Participants; unit: Participants]
  currently smoking | 4 | 3 | 1 | 8
  quit smoking | 7 | 2 | 2 | 11
  never smoked | 4 | 2 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Cough
Description: Number of coughs during procedure as defined by cough requiring stopping procedure or treatment by anesthesiologist with propofol or alfentanyl
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: coughs
Arm/Group | Topical Lidocaine | Nebuliser Solution | Atomizer Solution
Number analyzed (Participants) | 15 | 7 | 7
coughs | 1.20 (1.70) | 1.71 (1.60) | 1.00 (1.00)

2. Secondary Outcome: Number of Participants With Post-procedure Sore Throat
Description: sore throat was self reported by patient as: none, mild, moderate, severe
Time Frame: 1 day
Population: The analysis population does not include subjects who left clinic prior to collection of this data
Measure: Count of Participants; unit: Participants
Arm/Group | Topical Lidocaine | Nebuliser Solution | Atomizer Solution
Number analyzed (Participants) | 11 | 6 | 6
Participants
  none | 6 | 4 | 2
  mild | 4 | 0 | 3
  moderate | 1 | 2 | 1
  severe | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Post-Procedure Subjective Cough
Description: Subjective cough as described by patient as: none, mild, moderate, severe
Time Frame: 1 day
Population: The analysis population does not include subjects who left clinic prior to collection of this data.
Measure: Count of Participants; unit: Participants
Arm/Group | Topical Lidocaine | Nebuliser Solution | Atomizer Solution
Number analyzed (Participants) | 11 | 6 | 6
Participants
  none | 1 | 1 | 2
  mild | 8 | 4 | 3
  moderate | 2 | 1 | 1
  severe | 0 | 0 | 0

4. Secondary Outcome: Anesthesia Time to Wake up
Description: time in minutes from scope out until ready for transport to post anesthesia care unit
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Topical Lidocaine | Nebuliser Solution | Atomizer Solution
Number analyzed (Participants) | 15 | 7 | 7
minutes | 8.47 (4.02) | 13.00 (5.77) | 6.14 (3.80)

5. Secondary Outcome: Alfentanyl Dosing
Description: Total alfentanyl dosing by anesthesia in mcg/kg
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: mcg/kg
Arm/Group | Topical Lidocaine | Nebuliser Solution | Atomizer Solution
Number analyzed (Participants) | 15 | 7 | 7
mcg/kg | 16.61 (22.64) | 47.99 (37.41) | 4.40 (7.42)

6. Secondary Outcome: Propofol Dosing
Description: Total propofol dosing by anesthesia in mg/kg
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Topical Lidocaine | Nebuliser Solution | Atomizer Solution
Number analyzed (Participants) | 15 | 7 | 7
mg/kg | 5.30 (3.23) | 6.93 (3.36) | 3.26 (0.81)

7. Secondary Outcome: Fentanyl Dosing
Description: total fentanyl dosing by anesthesia in mcg/kg
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: mcg/kg
Arm/Group | Topical Lidocaine | Nebuliser Solution | Atomizer Solution
Number analyzed (Participants) | 15 | 7 | 7
mcg/kg | 0.30 (0.28) | 0.24 (0.23) | 0.48 (0.39)

ADVERSE EVENTS:
Time Frame: Data collected in the post-anesthesia care unit up to 1 hour after procedure
Arm/Group | Topical Lidocaine | Nebuliser Solution | Nebuliser Suspension
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/15 | 0/7 | 0/7

LIMITATIONS AND CAVEATS:
The target enrollment was not reached secondary to the COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-10): https://cdn.clinicaltrials.gov/large-docs/18/NCT03829618/Prot_SAP_000.pdf